CLINICAL TRIAL: NCT01632917
Title: Phase 1, Open-Label, Randomized, Safety and Pharmacokinetic Study of Two Final Formulations of ATX-101 (Sodium Deoxycholate Injection) Following Subcutaneous Injections in the Submental Fat
Brief Title: Open-Label Pharmacokinetic Study of Final Formulations of ATX-101
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kythera Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATX-101-12-32
Record Dates: First submitted 2012-06-29; First posted 2012-07-03 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Healthy
Keywords: Healthy volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ATX-101 - EU (Experimental): Open Label study in which subjects will receive ATX-101 (one of the two formulations) in one dosing session in the submental area
  Interventions: Drug: ATX-101 - EU
- ATX-101 - US (Experimental): Open Label study in which subjects will receive ATX-101 (one of the two formulations) in one dosing session in the submental area
  Interventions: Drug: ATX-101 - U.S.

INTERVENTIONS:
Drug: ATX-101 - U.S. — US ATX-101, 10 mg/mL, one dosing session in the submental area
  Arms: ATX-101 - US
Drug: ATX-101 - EU — EU ATX-101, 10 mg/mL, one dosing session in the submental area
  Arms: ATX-101 - EU

SUMMARY:
The objectives of this trial are to evaluate the safety and tolerability of ATX-101 injections and to characterize the pharmacokinetic profile of the two ATX-101 formulations.

DETAILED DESCRIPTION:
The objectives of this trial are to evaluate the safety and tolerability of ATX-101 injections and to characterize the pharmacokinetic profile of the two ATX-101 formulations that are expected to be the final formulations. ATX-101 will be administered into the submental fat as subcutaneous injections using the maximum proposed dosing regimen that is intended for labeling.

ELIGIBILITY:
Inclusion Criteria:

* Presence of sufficient submental fat into which 50 subcutaneous injections of ATX-101 spaced on a 1.0-cm grid can be safely administered based on the investigator's judgment.
* Males or nonpregnant, nonlactating females who are aged 18 to 65 years, inclusive, on the date of dosing with ATX-101. Females must have a negative serum human chorionic gonadotropin (hCG) test result from a sample obtained during the screening period and after admission to the research facility, but before the dose of study material. Females of postmenopausal status must not have had menses for at least one year and if younger than 55 years of age must have a serum FSH level ≥ 35 mIU/mL. Females of childbearing potential must agree to practice adequate contraception, in the judgment of the investigator, during the course of the trial.
* Serum hemoglobin test result of 11.0 g/dL or greater and negative hepatitis B, hepatitis C, and HIV test result within 28 days before the dose of study material.
* Willing and able to comply with and understand the visit schedule and all of the protocol-specified tests and procedures.
* Medically able to undergo the administration of study material as determined by clinical and laboratory evaluations obtained within 28 days before dosing with study material for which the investigator identifies no clinically significant abnormality.
* Signed informed consent obtained before any study-specific procedure is conducted.

Exclusion Criteria:

* History of any intervention to treat submental fat (e.g. liposuction, surgery, or lipolytic agents).
* History of trauma associated with the chin or neck areas, which in the judgment of the investigator may affect evaluation of safety of treatment.
* Loose skin in the neck or chin area for which reduction in submental fat may, in the judgment of the investigator, result in a cosmetically unacceptable outcome.
* Prominent platysmal bands at rest that interfere with the evaluation of submental fat.
* Evidence of any cause of enlargement in the submental area other than localized subcutaneous fat.
* Body mass index (BMI) > 40.0 at the screening visit. Refer to Appendix B.
* Use of tobacco or nicotine-containing products within 3 months prior to dose.
* Any blood donation or significant blood loss within 56 days before the dose of study material or plasma donation within 7 days before the dose of study material.
* A result on coagulation tests (PT, PTT) obtained within 28 days before the dose of study material that indicates the presence of any clinically significant bleeding disorder.
* Any medical condition that would interfere with the assessment of safety in this trial or would compromise the ability of the subject to undergo study procedures or to give informed consent.
* Treatment with fish oil, aspirin, or nonsteroidal anti-inflammatory agents (NSAIDS), except acetaminophen, within 7 days before dosing, or any anticipated need for agents with anticoagulative effects (e.g. warfarin, heparin) during the course of the trial.
* Treatment with oral anticoagulants (e.g. warfarin) within 30 days before dosing with study material.
* Treatment with radio frequency, laser procedures, chemical peels, or dermal fillers in the neck or chin area within 12 months before dosing with the study material, or botulinum toxin injections in the neck or chin area within 6 months before dosing with the study material.
* History of sensitivity to any components of the study material.
* History of drug or alcohol abuse, in the judgment of the investigator, within two years before dosing with the study material.
* Presence of a positive urine drug or alcohol screening test result obtained from a sample obtained during the screening period and/or after admission to the research facility for the confinement period, but before dosing with the study material.
* Previous enrollment into a trial of ATX-101.
* Treatment with an investigational device or agent within 30 days before dosing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Safety of ATX-101 injections as assessed by incidence, severity and duration of AEs of ATX-101 administered into subcutaneous fat in the submental and abdomen area | 8 days
  Spontaneously reported adverse events, laboratory test results, and treatment area evaluations including, but not limited to evaluation of edema, bruising, dysphagia, dysphonia, erythema, dyspigmentation, induration, numbness, pain, paresthesia, and pruritus.

SECONDARY OUTCOMES:
To compare the pharmacokinetic profile (Cmax, tmax, AUC, half-life) of ATX-101 administered into subcutaneous fat in the submental area | 8 days
  Blood sampling at specified time points before and after dosing with ATX-101 for analysis of deoxycholate concentrations in the plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Walker, MD, PhD, Study Director — Kythera Biopharmaceuticals, Inc
Locations (1):
- Comprehensive Clinical Development, Miramar, Florida, United States